CLINICAL TRIAL: NCT06751290
Title: The Use of Cyproheptadine to Improve Eating Habits in Children With Pediatric Feeding Disorders
Brief Title: The Use of Cyproheptadine in Pediatric Feeding Disorders
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Miguel Saps, Professor of Clinical, University of Miami
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20240756
Record Dates: First submitted 2024-10-31; First posted 2024-12-27 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Pediatric Feeding Disorder, Chronic; Avoidant Restrictive Food Intake Disorder
Keywords: Cyproheptadine; Malnutrition
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome; Avoidant Restrictive Food Intake Disorder; Malnutrition | interventions — Cyproheptadine; Nutrition Assessment; Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nutritional Counseling in Combination with Behavioral Counseling (Experimental): Participants in the group will receive nutritional and behavioral counseling for up to 6 months
  Interventions: Behavioral: Nutritional Counseling; Behavioral: Behavioral Counseling
- Cyproheptadine (Experimental): Participants in this group will receive the Cyproheptadine for up to 6 months
  Interventions: Drug: Cyproheptadine; Behavioral: Nutritional Counseling; Behavioral: Behavioral Counseling

INTERVENTIONS:
Drug: Cyproheptadine — Initiation of Cyproheptadine at 0.25mg/kg once daily by mouth at bedtime and titration up to at most three times daily as per participant's primary gastroenterologist.
  Arms: Cyproheptadine
Behavioral: Nutritional Counseling — This includes in person counseling by a provider once in office for up to 15 minutes as well as standardized hand out with basic nutritional guidance on high-calorie foods.
Behavioral: Behavioral Counseling — This includes in person counseling by a provider once in office for up to 15 minutes as well as standardized hand out with basic behavioral guidance.

SUMMARY:
The goal of this clinical trial is to learn if Cyproheptadine, an appetite stimulant, can improve eating habits in children with Pediatric Feeding Disorders. Pediatric Feeding Disorders is a broad term that describes disorders of eating-related behaviors that causes altered consumption of food and impairs physical or psychosocial health.

ELIGIBILITY:
Inclusion Criteria:

* Any patient aged 2-6 years of age who presents to Pediatric Gastroenterology Clinic with complaint of "poor weight gain, malnutrition, failure to thrive/weight faltering, picky eating, or feeding issues" who screens positive for a pediatric feeding disorder using the Child eating disorder questionnaire (CEBQ)
* Age Range: 2-6 years
* English or Spanish speaking

Exclusion Criteria:

* Patients who are tube fed
* Patients who are overweight (BMI at 85th%tile or greater)
* Patients who have active symptoms from a diagnosis of a GI disorder (Inflammatory Bowel Disease, Eosinophilic Esophagitis, Gastritis)
* Patients actively undergoing behavioral feeding therapy

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2024-12-30 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in Children's Eating Behavior Questionnaire score | Baseline and up to 6 months
  A composite score will be obtained and scores range from 1-5 with higher scores indicating more behavioral eating.
Number of foods consumed by participants | Baseline and up to 6 months
  Number of food consumed will be collected. Number of foods consumed as defined as eaten more than once per month.
Change in Child Food Neophobia score | Baseline and up to 6 months
  Score of 10-70 with higher score indicating higher neophobia.

SECONDARY OUTCOMES:
Change in weight | Baseline and up to 6 months
  Weight measured in kilograms
Change in height | Baseline and up to 6 months
  Height measured in centimeters
Change in BMI | Baseline and up to 6 months
  BMI measured in kg/m2
Change in BMI percentile | Baseline and up to 6 months
  BMI measured in percent
Change in BMI Z-score | Baseline and up to 6 months
  BMI measured in standard deviation units
Number of treatment related adverse events | Up to 6 months
  Number of treatment related adverse events using the National Cancer Institute (NCI) common terminology criteria for adverse events (CTCAE) version 5 as per physician discretion.
Parent's perception of medication's effects | Up to 6 months
  Measured by Cyproheptadine Survey given to parents in yes/no format. Total sum of yes and no answers will be collected.

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Saps, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami Department of Pediatric Gastroenterology, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No